CLINICAL TRIAL: NCT07251582
Title: A Prospective Study on the Effect of Infusion Timing of Immune Checkpoint Inhibitors on Pathologic Response in Patients With Resectable Stage II-III Non-Small Cell Lung Cancer Undergoing Neoadjuvant Therapy
Brief Title: Effect of Infusion Timing on Pathologic Response to Neoadjuvant Immunotherapy in Resectable Non-Small Cell Lung Cancer
Acronym: LungTime-C02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, DR, Hunan Province Tumor Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LungTime-C02
Record Dates: First submitted 2025-11-16; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Resectable Stage II-III Non-Small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; Time of day; neoadjuvant treatment
MeSH Terms: interventions — toripalimab; pembrolizumab; Platinum Compounds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning infusion group (Experimental): • Intervention / treatment:
  * Immune checkpoint inhibitor (one of approved PD 1 agents per investigator choice; e.g., toripalimab / pembrolizumab) administered in the morning window (08:00-11:00) for all ICI infusions during neoadjuvant treatment.
  * Combined with platinum based chemotherapy per institutional standard (examples: nab paclitaxel 260 mg/m² IV Day 1 Q3W + carboplatin AUC 5 IV Day 1 Q3W; or paclitaxel/cisplatin regimens per local practice).
  * Neoadjuvant treatment cycles: 4 cycles as per treating physician and local guideline; surgery scheduled after assessment.
  * Supportive care per routine practice.
  Interventions: Other: Time of Day-based Assignment for Infusion of Immune Checkpoint Inhibitor (e.g., toripalimab, or pembrolizumab) + platinum-based chemotherapy
- Afternoon infusion group (Active Comparator): • Intervention / treatment:
  * Same systemic regimen as Arm 1, but all ICI infusions administered in the afternoon window (15:00-18:00).
  * Chemotherapy, number of cycles (4), and surgical decision follow the same rules as Arm 1.
  * Supportive care per routine practice.
  Interventions: Other: Time of Day-based Assignment for Infusion of Immune Checkpoint Inhibitor (e.g., toripalimab, or pembrolizumab) + platinum-based chemotherapy

INTERVENTIONS:
Other: Time of Day-based Assignment for Infusion of Immune Checkpoint Inhibitor (e.g., toripalimab, or pembrolizumab) + platinum-based chemotherapy — Patients will be randomly assigned (1:1) to receive all ICI infusions during either the morning window (08:00-11:00) or the afternoon window (15:00-18:00), throughout the neoadjuvant treatment period.

SUMMARY:
This prospective study aims to investigate whether the time of day when immune checkpoint inhibitors (ICIs) are administered affects the efficacy of neoadjuvant immunotherapy in patients with resectable stage II-III non-small cell lung cancer (NSCLC). Eligible patients will receive standard-of-care neoadjuvant ICI plus platinum-based chemotherapy and be randomly assigned to either a morning infusion group (08:00-11:00) or an afternoon infusion group (15:00-18:00). The primary objective is to compare the pathological complete response (pCR) rates between groups. Secondary outcomes include major pathological response (MPR) and event-free survival (EFS). The study will include independent imaging and pathology review for endpoint assessment.

DETAILED DESCRIPTION:
Emerging evidence suggests that the efficacy of immune checkpoint inhibitors (ICIs) may be influenced by the circadian timing of drug administration. Retrospective studies in multiple cancer types have indicated that morning infusion of ICIs might be associated with improved clinical outcomes compared to afternoon infusion. However, no prospective study has evaluated this phenomenon in the setting of neoadjuvant therapy for resectable non-small cell lung cancer (NSCLC).

This prospective, randomized, parallel-group study aims to assess whether the time of day of ICI infusion (morning vs. afternoon) affects the pathological response to neoadjuvant immunotherapy in patients with stage II-III resectable NSCLC.

Eligible patients will receive standard-of-care neoadjuvant treatment, consisting of an immune checkpoint inhibitor (e.g., toripalimab, or pembrolizumab) combined with platinum-based chemotherapy. Patients will be randomly assigned (1:1) to receive all ICI infusions during either the morning window (08:00-11:00) or the afternoon window (15:00-18:00), throughout the neoadjuvant treatment period.

The primary endpoint is the pathological complete response (pCR) rate after neoadjuvant therapy and surgery. Secondary endpoints include major pathological response (MPR), event-free survival (EFS).The study will include independent imaging and pathology review for endpoint assessment.

This study aims to provide prospective evidence on the role of infusion timing in optimizing immunotherapy efficacy. If successful, this approach could offer a simple, cost-effective, and non-invasive strategy to improve outcomes for patients undergoing neoadjuvant immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

1. Age ≥18 and ≤75 years at the time of enrollment.
2. Histologically or cytologically confirmed diagnosis of resectable stage II to III non-small cell lung cancer (NSCLC).
3. Deemed suitable for neoadjuvant immunotherapy combined with platinum-based chemotherapy and subsequent surgical resection based on multidisciplinary team (MDT) assessment.
4. ECOG Performance Status of 0 or 1.
5. No prior systemic antitumor therapy for the current NSCLC diagnosis.
6. Adequate bone marrow, hepatic, renal, and cardiac function based on local laboratory standards.
7. Willing and able to comply with scheduled visits, treatment plans, and other study procedures.
8. Signed informed consent prior to participation.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded:

1. Presence of EGFR-sensitive mutations (e.g., exon 19del, L858R) or ALK/ROS1 rearrangements.
2. Presence of uncontrolled or symptomatic brain metastases.
3. History of any other malignancy within 3 years prior to enrollment, except for adequately treated basal cell carcinoma, squamous cell skin cancer, or cervical carcinoma in situ.
4. History of prior systemic therapy (immunotherapy, chemotherapy, or targeted therapy) for lung cancer.
5. Known severe allergic reactions to PD-1 or PD-L1 inhibitors (Grade ≥3 by CTCAE).
6. Active autoimmune disease requiring systemic immunosuppression.
7. Active infections, including active HBV, HCV, or HIV infection.
8. Pregnant or breastfeeding women.
9. Any comorbid condition or uncontrolled illness that, in the opinion of the investigator, may interfere with study participation or pose unacceptable risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-12-07 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate | At the time of surgery, approximately 6-9 weeks after randomization
  Proportion of patients achieving pathological complete response (no viable tumor cells in resected primary tumor and sampled regional lymph nodes) assessed on surgical specimen after completion of neoadjuvant therapy and surgery.

SECONDARY OUTCOMES:
Event Free Survival (EFS) | From date of randomization to event occurrence (disease progression, recurrence, or death), assessed up to 36 months
  Time from randomization to disease progression that precludes surgery, recurrence, or death from any cause, whichever occurs first.
Major Pathological Response (MPR) rate | At the time of surgery, approximately 6-9 weeks after randomization
  Proportion of patients with ≤10% viable tumor cells in the resected primary tumor specimen.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hunna Cancer Hospital, Clinical Trails Center, Changsha, Hunan
  - Hunan Cancer hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No